CLINICAL TRIAL: NCT01766102
Title: A Comparison of Intra-Operative Digital Specimen Mammography to Standard Specimen Mammography
Brief Title: Intra-operative Digital vs. Standard Mammography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michelle Specht, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-107
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- Intra-operative Mammography (Active Comparator): Intra-operative Specimen Mammography
  Interventions: Procedure: Intra-operative Mammography
- Standard Mammography (Active Comparator): Standard Specimen Mammography
  Interventions: Procedure: Standard Mammography

INTERVENTIONS:
Procedure: Intra-operative Mammography — The patient's breast specimen will be imaged in the operating room in an intra-operative imaging device - Biovision SN #30042
  Other Names: Biovision SN # 30042
  Arms: Intra-operative Mammography
Procedure: Standard Mammography — There is not an added device associated with this arm.
  Arms: Standard Mammography

SUMMARY:
A breast biopsy in the operating room may be needed in up to 15% of patients with an abnormality on mammogram. When an abnormality is present but there is no palpable mass, the abnormality must be localized with a wire before going to the operating room. This technique is also used when a breast cancer is present but there is no mass, in order to perform a targeted lumpectomy. Once the abnormality is surgically removed, the specimen with the wire is taken to the breast imaging department for a specimen x-ray to ensure that the targeted abnormality is present within the specimen. If the abnormality is close to the edge of the specimen, additional tissue is often removed.

A newer method for evaluating the specimen is to perform imaging in the operating room. Portable digital mammography units are available for this purpose. The Biovision digital specimen mammography system is FDA-approved and currently in use in over 200 centers in the United States. Several studies have shown that intra-operative digital mammography is as accurate as standard specimen mammography and takes less time to perform. It may also decrease the chance of having to go back to the operating room to take more breast tissue after lumpectomy because of cancer cells near teh margin(s) of the specimen on final pathology. Having to go back to the operating room to take more tissue is called a re-excision.

The purpose of this study is to compare standard specimen mammography to intra-operative specimen mammography to quantify potential operating room time savings and to determine if the use of intra-operative specimen mammography decreases re-excision rates. We aim to see if intra-operative specimen mammography is more efficient and if it decreases re-excision rates.

DETAILED DESCRIPTION:
Before the research starts patients will undergo some screening procedures to determine if patients are eligible to participate. This includes a medical history and an assessment of the patient's breast abnormality by mammogram and/or ultrasound and/or breast MRI. Patients will not need to undergo any extra procedures apart from those needed by the patient's surgeon to plan the patient's breast surgery. If the screening process shows that a patient is eligible to participate in this research study, the patient will be enrolled and the study will proceed on the day of surgery. If a patient does not meet the eligibility criteria the patient will not be able to participate in this research study.

Patients will be assigned to one of two arms of this study on the day of your surgery. Because no one knows which of the breast specimen imaging options is best, patients will be "randomized" into one of the study groups: the Standard Specimen Mammography arm or, the Intra-operative Specimen Mammography arm. Randomization means that the patient is put into a group by chance. It is like flipping a coin. Neither the patient nor the surgeon will choose what group the patient will be in.

If the patient is in the Standard Specimen Mammography arm, the patient's breast specimen (biopsy or lumpectomy) will be taken to the Breast Imaging department for a mammogram, which is the way breast specimens are typically imaged. If the patient is in the Intra-Operative Specimen Mammography arm, the patient's breast specimen will be imaged right in the operating room at the time of the surgery. The patient's images will also be linked to the Breast Imaging department, so the radiologist can confirm the surgeon's findings.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with a breast abnormality undergoing an excisional biopsy with wire localization or newly diagnosed with invasive breast cancer or ductal carcinoma undergoing a lumpectomy with wire localization
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Recurrent breast cancer
* Palpable masses not requiring wire localization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Specht, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intra-operative Mammography: Intra-operative Specimen Mammography
  Intra-operative Mammography: The patient's breast specimen will be imagine in the operating room in an intra-operative imaging device - Biovision SN #30042
Period: Overall Study
Arm/Group | Intra-operative Mammography | Standard Mammography
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-operative Mammography | Standard Mammography | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 79] | 57 [40 to 78] | 58 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 36 | 72
BMI [Median (Full Range); unit: Kg/m^2] — Body Mass Index is a weight to height ratio calculated by dividing someone's weight in Kg by the square of someone's height in meters.
  Kg/m^2 | 27 [18 to 38] | 25 [18 to 46] | 26 [18 to 46]
Reason for excision [Count of Participants; unit: Participants] — The indication for the excision:
  * An Excisional biopsy is a procedure where the entire abnormality or area of interest is removed.
  * Atypical Hyperplasia is a precancerous condition that is defined by an atypical accumulation of abnormal cells in the breast.
  * Ductal carcinoma in situ (DCIS) is the presence of abnormal cells inside a milk duct in the breast. DCIS is considered the earliest form of breast cancer.
  * Invasive Carcinoma is a cancer that began growing in a duct in the breast and has since invaded the fatty tissue of the breast outside of the duct.
  Participants
    Excisional Biopsy | 4 | 3 | 7
    Atypia | 7 | 5 | 12
    Invasive Carcinoma/DCIS | 25 | 28 | 53
Wire-localization Target [Count of Participants; unit: Participants] — A thin wire is inserted down to the target area of breast so that during surgery the surgeon can follow the guide wire down to the target area and remove the wire and the tissue around it. A clip is a marker that is placed in the breast during a biopsy that can be used a target for wire insertion. Mass means a solid mass in the breast. Calculated means that the target location was either manually or computer calculated. Architectural distortion (arch distort) is when a mammogram shows tethering or indentation of breast tissue but without an apparent associated mass.
  Participants
    Clip | 29 | 33 | 62
    Mass/ Calcs/ Arch distort | 7 | 3 | 10
Anesthesia Type [Count of Participants; unit: Participants] — The type of anesthesia used during the procedure. Monitored anesthesia care (MAC) is when a patient undergoes local anesthesia together with sedation and analgesia. General anesthesia is anesthesia that affects the whole body and usually induces a loss of consciousness.
  Participants
    MAC | 24 | 21 | 45
    General | 12 | 15 | 27
Axillary Surgery [Count of Participants; unit: Participants] — Type of axillary lymph node surgery
  * SLNB= Sentinel Lymph Node Biopsy
  * ALND= Axillary Lymph Node Dissection
  Participants
    None | 15 | 16 | 31
    SLNB | 20 | 20 | 40
    ALND | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Operative Time Savings
Description: To compare the overall operative time savings using intra-operative digital mammography compared with standard specimen mammography.
Time Frame: At the time of the procedure (approximately 1 week after randomization)
Measure: Median (Full Range); unit: Minutes
Arm/Group | Intra-operative Mammography | Standard Mammography
Number analyzed (Participants) | 36 | 36
Minutes
  Procedure Time | 48.5 [17 to 138] | 54 [17 to 140]
  OR Time | 68 [29 to 180] | 74 [35 to 177]
Statistical Analysis 1: Comparison: Intra-operative Mammography vs Standard Mammography; H0: Procedure time is not significantly different based on mammography type used; Test type: Other; p = 0.716, t-test, 2 sided
Statistical Analysis 2: Comparison: Intra-operative Mammography vs Standard Mammography; H0: Operating room time is not significantly different based on mammography type used; Test type: Other; p = 0.676, t-test, 2 sided

2. Secondary Outcome: Assessment of Radiographic and Pathologic Findings
Description: Assessment of radiographic findings and pathologic findings to determine sensitivity, specificity, positive predictive value, and negative predictive values of intra-operative digital specimen mammography (ISM) and standard specimen mammography for determining margin status.
  * A true positive (TP) was defined as a positive margin by imaging (ISM or SSM) and pathology
  * A false positive (FP) was defined as a positive margin by imaging but negative by pathology
  * A true negative (TN) was defined as a negative margin by both imaging and pathology.
  * A false negative (FN) was defined as a negative margin by imaging but positive by pathology
  * The sensitivity [TP/(TP + FN)], specificity [TN/(TN + FP)], positive predictive value [TP/ (TP + FP)], and negative predictive value [TN/(TN + FN)] for identification of positive margins were calculated for ISM and SSM.
Time Frame: 2 years
Population: Interpretation of margin status by the surgeon was available for 22 of 36 ISM patients. Interpretation of margin status was also available for 22 of 36 SSM patients.
Measure: Number; unit: Percent
Arm/Group | Intra-operative Mammography | Standard Mammography
Number analyzed (Participants) | 22 | 22
Percent
  Sensitivity | 50 | 20
  Specificity | 89 | 94
  Positive Predicitve Value | 50 | 50
  Negative Predictive Value | 89 | 80

ADVERSE EVENTS:
Description: Adverse Event information was not collected as a part of this trial
Arm/Group | Intra-operative Mammography | Standard Mammography
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes